CLINICAL TRIAL: NCT01970982
Title: A Controlled, 3-arm Parallel Group Study to Demonstrate Reduction in Exposure to Smoke Constituents in Healthy Smokers Switching to THS 2.2 or to Smoking Abstinence, Compared to Conventional Cigarettes for 5 Days in Confinement
Brief Title: Reduced Exposure Study in Smokers Using the Tobacco Heating System 2.2 (THS 2.2) for 5 Days in a Confinement Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZRHR-REXC-04-JP; ZRHR-REXC-04-JP (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2013-10-18; First posted 2013-10-28 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Candidate modified risk tobacco product; Conventional cigarette; Reduced exposure; HPHCs; Confinement
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tobacco Heating System (THS 2.2) (Experimental): Ad libitum use of THS 2.2 for 5 days in confinement
  Interventions: Other: Tobacco Heating System (THS 2.2)
- Smoking abstinence (SA) (Sham Comparator): Abstinence from smoking for 5 days in confinement
  Interventions: Other: Smoking abstinence (SA)
- Conventional cigarette (CC) (Active Comparator): Ad libitum use of Subject's own preferred brand of CC for 5 days in confinement
  Interventions: Other: Conventional cigarette (CC)

INTERVENTIONS:
Other: Tobacco Heating System (THS 2.2) — THS 2.2 ad libitum for 5 days in confinement
  Arms: Tobacco Heating System (THS 2.2)
Other: Smoking abstinence (SA) — SA for 5 days in confinement
  Arms: Smoking abstinence (SA)
Other: Conventional cigarette (CC) — Subject's own preferred brand of CC ad libitum for 5 days in confinement
  Arms: Conventional cigarette (CC)

SUMMARY:
The overall goal of the study is to evaluate if the ad libitum use of the Tobacco Heating System 2.2 (THS 2.2) for 5 consecutive days by adult Japanese healthy smokers affects the levels of biomarkers of exposure for selected harmful and potentially harmful constituents (HPHCs) compared to smoking conventional cigarettes (CC) and smoking abstinence (SA).

ELIGIBILITY:
Inclusion Criteria:

* Subject is Japanese.
* Smoking, healthy subject as judged by the Investigator.
* Subject smokes at least 10 commercially available non-menthol CCs per day (no brand restrictions) for the last 4 weeks, based on self reporting.
* Subject has smoked for at least the last 3 consecutive years.
* Subject does not plan to quit smoking in the next 3 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* The subject has received medication within 14 days or within 5 half-lives of the medication (whichever is longer), which has an impact on CYP1A2 or CYP2A6 activity.
* For women: Subject is pregnant or is breast feeding.
* For women: Subject does not agree to use an acceptable method of effective contraception.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takuya Kunito, MD, Principal Investigator — Higashi Shinjuku Clinic; Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (1):
- Higashi Shinjuku Clinic, Daito Building, 1-11-3, Okubo, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 23 July 2013
  At admission (Day -2), all the subjects performed a product trial of the THS 2.2. During the baseline period, they continued smoking their single preferred brand of CC. Then, on Day 0, subjects were randomized to one of the 3 study arms (THS 2.2, CC or SA) in a 2:1:1 ratio.
Pre-assignment Details: Enrolled and randomized population = 160 subjects
  * 80 subjects in THS 2.2
  * 40 subjects in CC
  * 40 subjects in SA
  Number of subjects enrolled but NOT randomized (who tried the THS 2.2 at Day -2) = 6
Period: Overall Study
Arm/Group | Tobacco Heating System (THS 2.2) | Conventional Cigarette (CC) | Smoking Abstinence (SA)
Started | 80 | 40 | 40
Completed | 80 | 40 | 38
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The study population consisted of all the randomized subjects who had at least 1 post randomization product use experience (THS 2.2 or CC arms), and 1 valid biomarker of exposure (BoExp) measurement.
  160 randomized subjects: 80 in THS 2.2, 40 in CC and 40 in SA
  158 completers: 2 subjects (SA arm) voluntarily withdrew on Day 1 and Day 3
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobacco Heating System (THS 2.2) | Conventional Cigarette (CC) | Smoking Abstinence (SA) | Total
Number analyzed (Participants) | 80 | 40 | 40 | 160
Age, Customized [Mean (Standard Deviation); unit: years]
  Between 23 and 65 years | 37.6 (11.7) | 37.2 (11.7) | 35.9 (10.6) | 37.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 20 | 80
  Male | 40 | 20 | 20 | 80
Daily CC consumption at Screening [Number; unit: participants]
  10 to 19 cig/day | 44 | 22 | 21 | 87
  > 19 cig/day | 36 | 18 | 19 | 73

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Monohydroxybutenyl Mercapturic Acid (MHBMA)
Description: Concentrations measured at Day 5 in urine, adjusted for creatinine.
  Geometric Least Squares LS) means are provided as descriptive statistics.
Time Frame: 5 days
Population: The analysis was performed on the full analysis set (FAS) population.
  The FAS consisted of all the randomized subjects who had at least 1 post randomization product use experience (if randomized to THS 2.2 or CC) and had at least 1 valid biomarker of exposure (BoExp) measurement (THS 2.2, CC, SA arms).
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | Tobacco Heating System (THS 2.2) | Conventional Cigarette (CC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 80 | 40 | 38
pg/mg creat | 106.25 [93.22 to 121.11] | 460.15 [382.54 to 553.51] | 91.73 [75.91 to 110.86]
Statistical Analysis 1: Comparison: Tobacco Heating System (THS 2.2) vs Conventional Cigarette (CC); The hypothesis to be tested is that the geometric mean level on Day 5 of the biomarker of exposure for THS 2.2 is lower relative to CC. Analysis of the BoExp was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 5 for THS 2.2 and CC respectively; Test type: Superiority or Other; p < 0.001, ANCOVA — The primary endpoints were tested using a multiple testing procedure to preserve the overall alpha level by simultaneously testing the endpoints using a closed procedure with each test performed at an alpha level of 2.5% one sided; ANCOVA model on MHBMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 23.09, 95% CI 2-sided [18.41 to 28.95] — LS mean ratio THS 2.2:CC

2. Primary Outcome: Concentration of 3-hydroxypropylmercapturic Acid (3-HPMA)
Description: Concentrations measured at Day 5 in urine, adjusted for creatinine.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 5 days
Population: The analysis was performed on the full analysis set (FAS) population.
  The FAS consisted of all the randomized subjects who had at least 1 post randomization product use experience (if randomized to THS 2.2 or CC) and had at least 1 valid BoExp measurement (THS 2.2, CC, SA arms).
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | Tobacco Heating System (THS 2.2) | Conventional Cigarette (CC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 80 | 40 | 38
ng/mg creat | 311.68 [286.43 to 339.16] | 589.65 [523.25 to 664.47] | 204.23 [180.70 to 230.82]
Statistical Analysis 1: Comparison: Tobacco Heating System (THS 2.2) vs Conventional Cigarette (CC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on 3-HPMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 52.86, 95% CI 2-sided [45.67 to 61.17] — LS mean ratio THS 2.2:CC

3. Primary Outcome: Concentration of S-phenylmercapturic Acid (S-PMA)
Description: as for outcome 2
Time Frame: 5 days
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | Tobacco Heating System (THS 2.2) | Conventional Cigarette (CC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 80 | 40 | 38
pg/mg creat | 142.05 [127.98 to 157.65] | 905.89 [781.81 to 1049.67] | 122.02 [104.92 to 141.90]
Statistical Analysis 1: Comparison: Tobacco Heating System (THS 2.2) vs Conventional Cigarette (CC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on S-PMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 15.68, 95% CI 2-sided [13.09 to 18.78] — LS mean ratio THS 2.2:CC

4. Primary Outcome: Levels of Carboxyhemoglobin (COHb)
Description: % COHb blood measurements performed in the evening of Day 5, expressed as % of saturation of hemoglobin.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 5 days
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: % of saturation of hemoglobin
Arm/Group | Tobacco Heating System (THS 2.2) | Conventional Cigarette (CC) | Smoking Abstinence (SA)
Number analyzed (Participants) | 80 | 40 | 38
% of saturation of hemoglobin | 2.41 [2.33 to 2.51] | 5.13 [4.87 to 5.39] | 2.37 [2.24 to 2.50]
Statistical Analysis 1: Comparison: Tobacco Heating System (THS 2.2) vs Conventional Cigarette (CC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on COHb levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 47.10, 95% CI 2-sided [44.30 to 50.08] — LS mean ratio THS 2.2:CC

ADVERSE EVENTS:
Time Frame: From the informed consent form (ICF) signature until the end of the safety follow-up period (7 days after discharge of the subject).
Description: The safety was assessed in the safety population, consisting of 166 subjects: 160 randomized subjects (80 in THS 2.2, 40 in CC and 40 in SA) and 6 subjects exposed to THS 2.2 from the product trial on Day -2 but not randomized.
Groups:
- Enrolled But Not Randomized: Subjects who tried the THS 2.2 at Admission (Day -2) but were not randomized in 1 of the 3 arms as they were back-up subjects
Arm/Group | Tobacco Heating System (THS 2.2) | Conventional Cigarette (CC) | Smoking Abstinence (SA) | Enrolled But Not Randomized
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/40 | 0/40 | 0/6
Other Adverse Events (participants affected / at risk) | 2/80 | 2/40 | 0/40 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tobacco Heating System (THS 2.2) (N=80) | Conventional Cigarette (CC) (N=40) | Smoking Abstinence (SA) (N=40) | Enrolled But Not Randomized (N=6)
Blood triglycerides increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belongs to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2013-07-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT01970982/Prot_000.pdf
  • Statistical Analysis Plan (2014-06-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT01970982/SAP_001.pdf